CLINICAL TRIAL: NCT02831283
Title: Imaging Inflammation in Elders With Different Clinical and Biomarker Profiles of Alzheimer's Disease
Brief Title: Imaging Inflammation in Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Patrick Lao (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Patrick Lao, Assistant Professor of Neurology, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAO1151; 1K23AG052633-01 (NIH)
Record Dates: First submitted 2016-07-10; First posted 2016-07-13 (Estimated); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer's Disease
Keywords: inflammation; aging; mild cognitive impairment
MeSH Terms: conditions — Alzheimer Disease; Inflammation; Cognitive Dysfunction | interventions — (methyl-(11)C)N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine; 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene; Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Amyloid-positive with cognitive impairment (AD) (Experimental): Amyloid-positive patients who already have cognitive impairment at the time of enrollment.
  Interventions: Drug: 11C-PBR28; Drug: 18F-Florbetaben; Procedure: Lumbar puncture (optional)
- Amyloid-positive without impairment (preclinical AD) (Active Comparator): Cognitively normal subjects who are amyloid-positive
  Interventions: Drug: 11C-PBR28; Drug: 18F-Florbetaben; Procedure: Lumbar puncture (optional)
- Amyloid-negative with cognitive impairment (Active Comparator): Participants with cognitive impairment due to suspected non-AD pathophysiology
  Interventions: Drug: 11C-PBR28; Drug: 18F-Florbetaben; Procedure: Lumbar puncture (optional)
- Amyloid-negative without impairment (normal aging) (Active Comparator): Cognitively normal subjects who are amyloid-negative on PET, and lack signs of neurodegeneration from other biomarkers
  Interventions: Drug: 11C-PBR28; Drug: 18F-Florbetaben; Procedure: Lumbar puncture (optional)

INTERVENTIONS:
Drug: 11C-PBR28 — 11C-PBR28 is a PET radioligand that binds to the 18 kDa translocator protein (TSPO), a marker of inflammation. 11C-PBR28 has previously been administered in humans. 11C-PBR28 will be administered at activity of up to 20 mCi per injection.
  Other Names: 11C-[O-methyl-11C]N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine
Drug: 18F-Florbetaben — 18F-Florbetaben (Neuraceq) has FDA approval for human use in evaluation of Alzheimer's disease. 18F-Florbetaben will be administered at activity up to 8.1 mCi per injection.
  Other Names: Neuraceq
Procedure: Lumbar puncture (optional) — Subjects have the option to have lumbar puncture performed for the measurement of inflammatory markers in cerebrospinal fluid.
  Other Names: LP

SUMMARY:
This study is being done to learn about inflammation and amyloid in Alzheimer's disease. A type of brain scan called a PET scan is used measure 1) inflammation and 2) abnormal accumulation of a the amount of a certain protein fragment called beta-amyloid (plaques) in the brain. These are thought to be involved in Alzheimer's disease. The investigators will also perform brain MRI and do tests to measure the participants' memory and thinking.

DETAILED DESCRIPTION:
This study is being done to determine the relationship between inflammation, cognitive impairment, and amyloid burden in elderly subjects with different clinical and biomarker profiles of Alzheimer's disease (AD). Participants will undergo amyloid PET imaging with 18F-Florbetaben with target number of completers being 15 amyloid-positive elders with impairment, 15 amyloid-positive elders with normal cognition, 15 amyloid-negative elders with impairment, and 15 amyloid-negative elders with normal cognition. Subjects will undergo screen that includes neuropsychological testing, brain MRI, and PET imaging with 18F-florbetaben to define the above 4 groups. Subjects will have 11C-PBR28 PET imaging to measure the 18 kDa translocator protein (a marker of inflammation). Subjects will have the option to have lumbar puncture performed to measure CSF concentrations of amyloid,tau, phospho-tau, and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 and older.
2. Meet criteria for either a) amnestic mild cognitive impairment (single or mixed domain) or mild Alzheimer's disease, or b) have no cognitive impairment based on history, exam, neuropsychological testing, and consensus diagnosis. MCI and mild AD patients must have Clinical Dementia Rating scale score of 0.5 or 1. Unimpaired subjects must have Clinical Dementia Rating scale score of 0.
3. Subjects unable to provide informed consent must have a surrogate decision maker
4. Written and oral fluency in English or Spanish.
5. Able to participate in all scheduled evaluations and to complete all required tests and procedures.
6. In the opinion of the investigator, the subject must be considered likely to comply with the study protocol and to have a high probability of completing the study.

Exclusion Criteria:

1. Past or present history of certain brain disorders other than MCI or AD.
2. Certain significant medical conditions, which make study procedures of the current study unsafe.
3. Contraindication to MRI scanning.
4. Conditions precluding entry into the scanners (e.g., morbid obesity, claustrophobia, etc.).
5. Exposure to research related radiation in the past year that, when combined with this study, would place subjects above the allowable limits.
6. Low affinity binding on TSPO genetic screen.
7. Participation in the last year in a clinical trial for a disease modifying drug for AD.
8. Inability to have a catheter in subject's vein for the injection of radioligand.
9. Inability to have blood drawn from subject's veins.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06; Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Lao, Principal Investigator — Columbia University
Locations (1):
- Columbia University irving Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Klein J, Yan X, Johnson A, Tomljanovic Z, Zou J, Polly K, Honig LS, Brickman AM, Stern Y, Devanand DP, Lee S, Kreisl WC. Olfactory Impairment Is Related to Tau Pathology and Neuroinflammation in Alzheimer's Disease. J Alzheimers Dis. 2021;80(3):1051-1065. doi: 10.3233/JAD-201149. PMID 33646153

RESULTS

PARTICIPANT FLOW:
Groups:
- Amyloid-negative Without Impairment (Normal Aging): Cognitively normal subjects who are amyloid-negative on PET and lack signs of neurodegeneration from other biomarkers
Period: Overall Study
Arm/Group | Amyloid-positive With Cognitive Impairment (AD) | Amyloid-positive Without Impairment (Preclinical AD) | Amyloid-negative With Cognitive Impairment | Amyloid-negative Without Impairment (Normal Aging)
Started | 24 | 8 | 11 | 17
Completed | 24 | 8 | 11 | 17
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amyloid-positive With Cognitive Impairment (AD) | Amyloid-positive Without Impairment (Preclinical AD) | Amyloid-negative With Cognitive Impairment | Amyloid-negative Without Impairment (Normal Aging) | Total
Number analyzed (Participants) | 24 | 8 | 11 | 17 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (8.7) | 73.8 (3.1) | 75.8 (9.8) | 67.6 (3.8) | 68.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 7 | 5 | 20
  Male | 20 | 4 | 4 | 12 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 1 | 2 | 6
  Not Hispanic or Latino | 21 | 8 | 10 | 15 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 6 | 9
  White | 24 | 6 | 10 | 11 | 51
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 11C-PBR28 Binding
Description: In vivo quantification radioligand binding to TSPO expression on microglia in the brain, reported as standardized uptake value ratio (SUVR).
Time Frame: Up to 1 year from screening
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Amyloid-positive With Cognitive Impairment (AD) | Amyloid-positive Without Impairment (Preclinical AD) | Amyloid-negative With Cognitive Impairment | Amyloid-negative Without Impairment (Normal Aging)
Number analyzed (Participants) | 24 | 8 | 11 | 17
SUVR | 1.25 (0.18) | 1.15 (0.16) | 1.16 (0.16) | 1.02 (0.13)

2. Secondary Outcome: 18F-Florbetaben Binding
Description: In vivo quantification of radioligand binding to Amyloid-Beta protein in the brain, reported as standardized uptake value ratio (SUVR).
Time Frame: Up to 1 year from screening
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Amyloid-positive With Cognitive Impairment (AD) | Amyloid-positive Without Impairment (Preclinical AD) | Amyloid-negative With Cognitive Impairment | Amyloid-negative Without Impairment (Normal Aging)
Number analyzed (Participants) | 24 | 8 | 11 | 17
SUVR | 1.64 (0.18) | 1.51 (0.14) | 1.17 (0.14) | 1.12 (0.06)

3. Secondary Outcome: Cerebral Spinal Fluid (CSF) Biomarkers
Description: Protein analysis of cerebral spinal fluid.
Time Frame: Up to 1 year from screening
Population: Some participants did not wish to do this procedure, so data was not collected from these participants.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Amyloid-positive With Cognitive Impairment (AD) | Amyloid-positive Without Impairment (Preclinical AD) | Amyloid-negative With Cognitive Impairment | Amyloid-negative Without Impairment (Normal Aging)
Number analyzed (Participants) | 12 | 4 | 3 | 5
ng/mL | 3.14 (1.69) | 4.21 (1.74) | 3.26 (2.99) | 2.05 (0.57)

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Amyloid-positive With Cognitive Impairment (AD) | Amyloid-positive Without Impairment (Preclinical AD) | Amyloid-negative With Cognitive Impairment | Amyloid-negative Without Impairment (Normal Aging)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/8 | 0/11 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/8 | 0/11 | 0/17
Other Adverse Events (participants affected / at risk) | 0/24 | 0/8 | 0/11 | 2/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amyloid-positive With Cognitive Impairment (AD) (N=24) | Amyloid-positive Without Impairment (Preclinical AD) (N=8) | Amyloid-negative With Cognitive Impairment (N=11) | Amyloid-negative Without Impairment (Normal Aging) (N=17)
Soreness at IV injection site (General disorders) | 0 | 0 | 0 | 1
Headache (General disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT02831283/Prot_SAP_000.pdf